CLINICAL TRIAL: NCT01507090
Title: Taking the Guesswork Out of Pediatric Weight Estimation (TAPE): Validation of the Mercy TAPE
Brief Title: Validation of the Mercy TAPE
Acronym: TAPE
Status: Completed | Type: Observational
Sponsor: Susan Abdel-Rahman (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Susan Abdel-Rahman, Professor of Pediatrics, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: Mercy TAPE
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Weight
Keywords: children for whom there is no scale to determine weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Children: Otherwise healthy children 2 months to 16 years of age.
  Interventions: Device: Mercy TAPE

INTERVENTIONS:
Device: Mercy TAPE — 2D Mercy TAPE and 3D Mercy TAPE

SUMMARY:
In 'real-world' health care settings there exist a number of circumstances where the weight of a child is desirable or even necessary but unavailable. Numerous weight estimation strategies have been described but each has limitations. Investigators at Children's Mercy Hospitals and Clinics recently developed a weight estimation method and tool that addresses the limitations of previously published methods. This study is intended to validate the device in a population of children 2 months to 16 years of age.

DETAILED DESCRIPTION:
In 'real-world' health care settings there exist a number of circumstances where the weight of a child is desirable or even necessary but unavailable. The most conspicuous of these settings can be found in developing countries where many medical clinics lack suitable scales to obtain accurate infant and child weights. Though resource restrictions are less of an issue in developed countries, scenarios still exist where weight assessment is problematic. For example, accurate estimates of a child's weight are rarely available during emergency or trauma situations, and in some in-patient settings (e.g. critical care units, orthopedic clinics) obtaining an accurate patient weight can be impaired by the presence of external hoses, tubing, casts, and/or other medical equipment. Irrespective of the environment, the challenge that each of these settings present is the same; namely, the provision of age-appropriate, weight-based interventions which remain the most accurate approach to delivering therapy in children. Thus, techniques which permit accurate weight estimation address a critical medical need in both developing and developed countries.

Numerous weight estimation strategies have been described with each used to varying degrees in clinical practice. Many of the published techniques have distinct advantages. For example; simple age-based equations can be used without the need for reference materials, strategies that utilize preprinted tables or tools limit the risk of calculation errors. Other techniques present unnecessary complexities for the end-user including; the need for subjective assessments of habitus, the requirement to solve exponential equations, the call for multiple formulae delineated by age bracket, or the reliance on one or more reference charts. Irrespective of their simplicity or complexity, almost all of the reported techniques have significant limitations. Relatively few methods have been evaluated in pediatric populations of varying races, ethnicities and nationalities and essentially no single previously described method provides accurate estimates of weight across broad age- and weight-bands.

Apart from parental recall which can vary in accuracy, the most commonly used strategies for estimating weight rely on the child's age, length, or a combination of the two parameters. While simple and easy to integrate into a weight estimation technique, age based strategies fail to account for the extremes of body composition and stature that are observed in children of the same age. Similarly, length based strategies do not take into consideration that two children of the same height may demonstrate markedly discrepant weights based on underlying nutritional status (e.g. malnourished, underweight, overweight, obese). Consequently, many of the currently available weight estimation strategies perform well in only a small subset of children. As such, there remains a critical need for weight estimation methods that are accurate across a wide range of pediatric ages, weights, lengths, nationalities and body compositions despite the relative abundance of strategies that already exist.

Investigators at Children's Mercy Hospitals and Clinics recently developed and validated a weight estimation method (the Mercy MethodTM) that addresses the principal limitations of previously published methods, requires no subjective assessment and performs robustly independently of age and length over a broad range of weights. As with other strategies, the Mercy Method incorporates growth velocity but uses humeral length as a surrogate for total body length. Total body length will be discrepant depending on whether the measurement is obtained with the child standing or lying down and can be difficult to obtain in a child who is uncooperative or obtunded. The Mercy Method also incorporates body habitus as a quantitative variable which improves the accuracy of the overall length-based weight estimate and removes the subjective nature of categorizing the child's body type into one of a few alternatives (e.g. "slim," "average," or "heavy"). By developing a model with these considerations in mind we were able to expand the age range to which our weight estimation method can be applied and remove length restrictions which are typically imposed because of the disproportionate increase in weight-for-height observed as children get older.

In brief, demographic and anthropometric data on children 2 months to 16 years of age were extracted from the NHANES database and individual datasets were randomly assigned into a method development (n=17,328) or a method validation (n=1,938) set. Humeral length (HL) and mid-upper arm circumference (MUAC) were used to develop a weight estimation method by 1) collapsing length and habitus measurements into discrete bins, 2) examining the median population weight for each bin-pair, 3) statistically weighting the bin-pairs for age and sample size, and 4) calculating a fractional weight for each HL and MUAC. An individual weight estimate is generated by the simple addition of the MUAC and HL fractional bin value that corresponds to that individual child's measurements. The predictive performance this method was evaluated using the internal validation set and compared with the performance of 13 previously published weight estimation methods applied to the same data.

The Mercy Method outperformed the 13 other published methods when evaluated for goodness-of-fit, mean error, mean percentage error, root mean square error and percentage of children in agreement within 10% of actual weight. Most of the age-and length-based strategies examined overestimated weight in children classified, by BMI, as underweight and significantly underestimated weight in children classified as overweight or obese. The degree to which this occurred depended largely on the constants driving their mathematical equations, with some methods biased toward more accurate prediction in children of lower weight (e.g. Broselow) and others performing better among children in the higher weight brackets (e.g. Theron). Irrespective of directionality, the bias observed with some methods at the extremes of weight represented as much as a 3-fold error between predicted and actual weights. Discrepancies of this magnitude can be dangerous, and potentially life-threatening, depending on how 'forgiving' the intervention or treatment that is being administered.

The singular habitus-based method (i.e. Cattermole) ranked among the best (after the Mercy Method) with respect to absolute bias; however, it performed only moderately well when precision and MPE were factored into the assessment. This method, which was developed in Chinese children consistently overestimated weight at lower absolute weights and underestimated weight at higher absolute weight irrespective of BMI percentile. This suggests that while the relationship between weight and MUAC tends to be linear within any given population, the mathematical constants that define the relationship differ between populations having different height-for-weight averages. Given the nature of the data used to develop and validate the Mercy Method, comparative performance of the Devised Weight Estimation Method (DWEM, the only other method to incorporate both body length and body habitus) could not be assessed. Notably, the DWEM involves a subjective rating of "slim," "average," or "heavy". While DWEM has been shown to outperform other age-based methods, the categorical assignment of habitus coupled with inconsistencies in subjective assessment between and within observers [inter-rater agreement- 78% (range: 58-93%); intra-rater agreement- 86% (range: 81-94%)] contributed to bias and precision estimates that were larger than observed with strategies based solely on length.

While the Mercy Method can be used as a reference table, a more practical application was the development of a simple and inexpensive device that can perform the two required measurements simultaneously and report the predicted weight directly from the device as opposed to consulting a separate table or chart. Consequently, the 3D Mercy TAPE was developed to perform both measurements simultaneously requiring no external references to arrive at the weight estimate for a given child. An alternative 2D Mercy TAPE was also designed . It requires two serial measurements with the same simple addition used with the 3D TAPE but does not require any folding or manipulation when removed from its packaging. Both devices are intended to be printed on any flexible, non-stretchable medium (e.g. paper, plastic coated paper, fiberglass) so as to be disposable or semi-permanent, inexpensive to mass produce and easy to store.

In its numeric form, the Mercy TAPE would be expected have limited utility in settings where care providers are illiterate or do not use a written language. However, the tool can be easily revised with colors and/or symbols whose combination would correspond to a given dose, intervention strategy or weight target. While the Mercy Method is expected to perform well in U.S. children given its creation using data from a U.S. database, external validation of the in non-U.S. settings is currently ongoing with support of the World Health Organization to gauge its utility in children of varying ethnicity and geographic origin. The related 2D and 3D Mercy TAPE still awaits prospective evaluation. The requisite study to satisfy the validation requirements are described herein under the hypothesis: The Mercy TAPE will demonstrate the same predictive performance as the Mercy method in an independent pediatric assessment.

ELIGIBILITY:
Inclusion Criteria:

* age between 2 months and 16 years of age
* capable of having the measurements performed
* parent or legal guardian is willing and able to provide verbal permission and, when appropriate, the participant has provided verbal assent to participate.

Exclusion Criteria:

* unwilling to participate in the study procedures
* known or apparent limb deformities
* presence of any external medical equipment attached to the child
* underlying pathological condition that would produce abnormal body composition for age (e.g. edema)
* underlying pharmacologic management that would produce abnormal body composition for age (e.g. chronic oral corticosteroid use)
* In the opinion of the physicians providing patient care and those conducting the study, there are real or perceived contraindications for inclusion as a participant in the study

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Normal healthy children
Sampling Method: Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Abdel-Rahman, Pharm.D, Principal Investigator — Childrens Mercy Hospital
Locations (3):
- United States (3):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Milton Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Derived] Abdel-Rahman SM, Paul IM, James LP, Lewandowski A; Best Pharmaceuticals for Children Act-Pediatric Trials Network. Evaluation of the Mercy TAPE: performance against the standard for pediatric weight estimation. Ann Emerg Med. 2013 Oct;62(4):332-339.e6. doi: 10.1016/j.annemergmed.2013.02.021. Epub 2013 Apr 17. PMID 23602655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from clinics, inpatient wards and referrals.
Groups:
- Normal Children: Otherwise healthy children 2 months to 16 years of age were enrolled. The 2D and 3D Mercy TAPE was developed to measure two upper arm landmarks so as to arrive at the weight estimate for a given child. The 2D Mercy TAPE requires two serial measurements with simple addition. The 3D TAPE makes both measurements simultaneously also requiring simple addition.
Period: Overall Study
Arm/Group | Normal Children
Started | 642
Completed | 624
Not Completed | 18
Not completed — incomplete dataset | 18

BASELINE CHARACTERISTICS:
Arm/Group | Normal Children
Number analyzed (Participants) | 642
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 642
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51.7
  Male | 48.3
Region of Enrollment [Number; unit: participants]
  United States | 642

OUTCOME MEASURES:

1. Primary Outcome: Predictive Performance of the Mercy TAPE (Percent of Participants Predicted Within 20% of Their Actual Weight)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with the actual weight (kg). Outcome measures reported below reflect the percentage of participants whose weight estimations using the Mercy TAPEs are within 20% of their actual weight.
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 2D-TAPE; 3D-TAPE: Otherwise healthy children 2 months to 16 years of age.
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
percentage of participants | 98.1 [97.0 to 99.2] | 93.3 [91.3 to 95.2]

2. Primary Outcome: Predictive Performance of the Mercy TAPE (Slope)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with the actual weight (kg). Outcome measures reported below reflect the slope of the regression equation comparing observed vs. predicted weight.
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
unitless | 0.980 [0.969 to 0.992] | 0.977 [0.964 to 0.990]

3. Secondary Outcome: Inter-rater Reliability for the 2D and 3D Mercy TAPEs.
Description: Intraclass correlation coefficient
Time Frame: study day 1
Population: All pre-qualified study coordinators
Measure: Number; unit: Intraclass correlation coefficient
Groups:
- 2D-TAPE; 3D-TAPE; Mercy Method: Study coordinators performing measurements
Arm/Group | 2D-TAPE | 3D-TAPE | Mercy Method
Number analyzed (Participants) | 16 | 16 | 16
Intraclass correlation coefficient | 0.993 | 0.980 | 0.990

4. Primary Outcome: Predictive Performance of the Mercy TAPE (Intercept)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with the actual weight (kg). Outcome measures reported below reflect the intercept of the regression equation comparing observed vs. predicted weight.
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number (95% Confidence Interval); unit: kilograms
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
kilograms | 0.968 [0.498 to 1.439] | 1.019 [0.464 to 1.573]

5. Primary Outcome: Predictive Performance of the Mercy TAPE (Mean Error)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
kilograms | 0.28 (3.3) | 0.22 (3.9)

6. Primary Outcome: Predictive Performance of the Mercy TAPE (Mean Percentage Error)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis
Measure: Mean (Standard Deviation); unit: percentage error
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
percentage error | 1.65 (8.5) | 1.91 (11.1)

7. Secondary Outcome: Device Print Batch Variability
Description: Geometric mean of the ratio (CV) of true to estimated weight calculated by TAPE version. Mercy TAPEs were printed in 2 batches numbers "1" and "2" accordingly.
Time Frame: study day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
ratio
  version 1 | 1.01 (0.08) | 1.02 (0.11)
  version 2 | 1.01 (0.09) | 1.01 (0.11)

8. Secondary Outcome: Predictive Performance of the Mercy Method (Intercept)
Description: Evaluate the weight generated by the Mercy method (kg) with the actual weight (kg)
Time Frame: study day 1
Measure: Number (95% Confidence Interval); unit: kilograms
Arm/Group | Normal Children
Number analyzed (Participants) | 624
kilograms | 1.083 [0.584 to 1.581]

9. Secondary Outcome: Predictive Performance of the Mercy Method (Slope)
Description: Evaluate the weight generated by the Mercy method (kg) with the actual weight (kg)
Time Frame: study day 1
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | Normal Children
Number analyzed (Participants) | 624
unitless | 0.980 [0.968 to 0.992]

10. Secondary Outcome: Predictive Performance of the Mercy Method (Percent of Participants)
Description: Evaluate the weight generated by the Mercy method (kg) with the actual weight (kg). The outcome measure below relfects the percent of participants with weight estimated within within 20% of actual weight.
Time Frame: study day 1
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Normal Children
Number analyzed (Participants) | 624
percent of participants | 97.3 [96.0 to 98.6]

11. Secondary Outcome: Predictive Performance of the Mercy Method (Mean Error)
Description: Evaluate the weight generated by the Mercy method (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Normal Children
Number analyzed (Participants) | 624
kilograms | 0.39 (3.5)

12. Primary Outcome: Predictive Performance of the Mercy TAPE (Corelation Coefficient)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis
Measure: Number; unit: correlation coefficient
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
correlation coefficient | 0.979 | 0.971

13. Primary Outcome: Predictive Performance of the Mercy TAPE
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis
Measure: Number; unit: root mean square error (kg)
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
root mean square error (kg) | 3.33 | 3.92

14. Primary Outcome: Equivalence of the Mercy Method and the 2D and 3D Mercy TAPEs (Ratio)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with weight generated by the Mercy method (kg). Outcome measures reported below reflect the slope of the regression equation comparing method predicted vs. TAPE predicted weight.
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
unitless | 0.998 [0.994 to 1.002] | 0.998 [0.991 to 1.005]

15. Primary Outcome: Equivalence of the Mercy Method and the 2D and 3D Mercy TAPEs (Concordance Corelation Coefficient)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with weight generated by the Mercy method (kg). Outcome measures reported below reflect the intercept of the regression equation comparing method predicted vs. TAPE predicted weight.
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
unitless | 0.996 [0.996 to 0.997] | 0.993 [0.991 to 0.994]

16. Primary Outcome: Equivalence of the Mercy Method and the 2D and 3D Mercy TAPEs (% Within 10%)
Description: Evaluate the weight generated by the 2D and 3D Mercy TAPE (kg) with weight generated by the Mercy method (kg). Outcome measures reported below reflect the percentage weight estimations using the Mercy TAPEs that are within 10% of the weight estimations using the Mercy Method.
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number (95% Confidence Interval); unit: percent of estimations
Arm/Group | 2D-TAPE | 3D-TAPE
Number analyzed (Participants) | 624 | 624
percent of estimations | 91.7 [89.5 to 93.8] | 76.4 [73.1 to 79.8]

17. Secondary Outcome: Predictive Performance of the Mercy Method (Mean Percentage Error)
Description: Evaluate the weight generated by the Mercy method (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Mean (Standard Deviation); unit: percentage error
Arm/Group | Normal Children
Number analyzed (Participants) | 624
percentage error | 1.86 (8.9)

18. Secondary Outcome: Predictive Performance of the Mercy Method
Description: Evaluate the weight generated by the Mercy method (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number; unit: correlation coefficieint
Arm/Group | Normal Children
Number analyzed (Participants) | 624
correlation coefficieint | 0.977

19. Secondary Outcome: Predictive Performance of the Mercy Method
Description: Evaluate the weight generated by the Mercy method (kg) with the actual weight (kg)
Time Frame: study day 1
Population: Final population for data analysis.
Measure: Number; unit: root mean square error (kg)
Arm/Group | Normal Children
Number analyzed (Participants) | 624
root mean square error (kg) | 3.55

ADVERSE EVENTS:
Description: For the purpose of this study, only adverse events and serious adverse events directly associated to the measurement procedures were assessed. Adverse event reporting ocuured within a 20 minute window of the measurement procedure.
Arm/Group | Normal Children
Serious Adverse Events (participants affected / at risk) | 0/642
Other Adverse Events (participants affected / at risk) | 0/642

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes